CLINICAL TRIAL: NCT00154388
Title: Phase II Study of Imatinib Mesylate in Patients With Life Threatening Malignant Rare Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571B2225
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Life Threatening Diseases
Keywords: adenocarcinoma; leiomyosarcoma; angiosarcoma; synovial sarcoma; myelodysplastic syndrome/HES; CMML; multiple myeloma; embryonal rhabdomyosarcoma; endometrial sarcoma; adenoid cystic carcinoma; fibromatosis; ductal invasive breast carcinoma; chondrosarcoma; pleural tumor; brenner tumor; ewing sarcoma; round cell tumor; seminoma; thymic carcinoma; malignant melanoma; fibrosarcoma breast; dermatofibrosarcoma protuberans; DFSP; ovarian stromal tumor; osteosarcoma; chorioideal melanoma; hemangiopericytoma; myelofibrosis; liposarcoma; SCLC; small cell lung carcinoma; hypereosinophilic syndrome; chronic myelo-monocytic leukemia; neurofibrosarcoma; mesothelioma; malignant mesenchymoma; malignant schwannoma; mast cell leukemia / mastocytosis; renal cell carcinoma; malignant histocytoma; chordoma
MeSH Terms: conditions — Adenocarcinoma; Leiomyosarcoma; Hemangiosarcoma; Sarcoma, Synovial; Multiple Myeloma; Rhabdomyosarcoma, Embryonal; Sarcoma, Endometrial Stromal; Carcinoma, Adenoid Cystic; Fibroma; Carcinoma, Ductal, Breast; Chondrosarcoma; Pleural Neoplasms; Brenner Tumor; Sarcoma, Ewing; Seminoma; Thymoma; Melanoma; Dermatofibrosarcoma; Osteosarcoma; Hemangiopericytoma; Primary Myelofibrosis; Liposarcoma; Small Cell Lung Carcinoma; Hypereosinophilic Syndrome; Neurofibrosarcoma; Mesothelioma; Malignant mesenchymal tumor; Leukemia, Mast-Cell; Mastocytosis; Carcinoma, Renal Cell; Chordoma | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib mesylate

SUMMARY:
Exploratory study to examine the effect(s) of Imatinib mesylate treatment on life threatening rare diseases with known associations to one or more Imatinib mesylate -sensitive tyrosine kinases, and to identify the contribution of specific protein tyrosine kinases (PTKs) of that specific disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 15 years of age
* Life threatening disease documented by conventional criteria to be resistant to standard, approved therapy.
* Experimental documentation of functional significance of either Abl, Kit (CD117), or PDGF-R in the relevant target tissue (preferably on a sample taken within 6 weeks of study entry).
* ECOG Performance status of 0, 1, or 2.
* Adequate end organ function defined as: total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL (or < 5 x ULN for patients with hepatic disease), creatinine < 1.5 x ULN, ANC > 1.5 x 109/L, platelets > 100 x 109/L.
* Negative serum or urine pregnancy test for women of child bearing potential (WOCBP) within 7 days of study initiation. Post menopausal women must have experienced amenorrhea for at least 12 months. Male and female patients must use effective birth control methods throughout the study and for up to 3 months after study discontinuation.
* Life expectancy of more than 3 months.
* Written, voluntary, informed consent for retrieval, evaluation and investigational use of tissue samples.

Exclusion Criteria:

* Patients who have received any other investigational agent within 28 days of study initiation.
* Patients with another primary malignancy except if other primary malignancy is neither currently clinically significant nor requiring active intervention.
* Patients with Grade III/IV cardiac problems defined by the New York Heart Association Criteria (e.g. congestive heart failure, myocardial infarction within 6 months of study).
* Female patients who are pregnant or breast-feeding.
* Patients who have another severe and/or life threatening medical disease.
* Patients with acute or known chronic liver disease (e.g. chronic active hepatitis, cirrhosis).
* Patients with a known diagnosis of the human immunodeficiency virus ((HIV) infection.
* Patients who have received chemotherapy within 4 weeks (6 weeks allowed for nitrosourea, mitomycin-C or any antibody therapy) prior to study entry.
* Patients who have had major surgery within 2 weeks prior to study entry.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2001-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To examine the effect(s) of Imatinib mesylate treatment on life threatening rare diseases with known associations to one or more Imatinib mesylate-sensitive tyrosine kinases
To identify the contribution of specific protein tyrosine kinases (PTKs) of that specific disease

SECONDARY OUTCOMES:
To assess the safety and tolerability of Imatinib mesylate
To evaluate the pharmacokinetic profile of Imatinib mesylate
To assess, where feasible, the functional significance of relevant signal-transduction components in target tissues

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heinrich, MD, Principal Investigator — Oregon Health and Science University

REFERENCES:
- [Result] Chugh R, Wathen JK, Maki RG, Benjamin RS, Patel SR, Meyers PA, Priebat DA, Reinke DK, Thomas DG, Keohan ML, Samuels BL, Baker LH. Phase II multicenter trial of imatinib in 10 histologic subtypes of sarcoma using a bayesian hierarchical statistical model. J Clin Oncol. 2009 Jul 1;27(19):3148-53. doi: 10.1200/JCO.2008.20.5054. Epub 2009 May 18. PMID 19451433